CLINICAL TRIAL: NCT04150757
Title: The Use of Intranasal (IN) Ketamine for Pain Control in Patients with Sickle Cell Disease and Vaso-occlusive Episode (VOE) in the Pediatric Emergency Department
Brief Title: Intranasal Ketamine for Pain Control in Patients with Sickle Cell Disease and Vaso-occlusive Episode (VOE) in the PED
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment secondary to COVID
Sponsor: Abigail Nixon (Other)
Responsible Party: Sponsor-Investigator, Abigail Nixon, Principle Investigator, MD, New York City Health and Hospitals Corporation
Organization: New York City Health and Hospitals Corporation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10379
Record Dates: First submitted 2019-10-16; First posted 2019-11-05 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease; Vaso-Occlusive Pain Episode in Sickle Cell Disease; Vaso-occlusive Crisis; Ketamine; Intranasal Ketamine; Analgesia
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Agnosia

STUDY DESIGN:
Intervention Model Description: Enrolled patients will receive one dose of Intranasal Ketamine dosed at 1mg/kg (Ketamine 500mg/10 mL solution) after triage while waiting for IV placement (max 50mg). This is an observational study.
Masking Description: Patients and treating providers will be aware of the medication administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Analgesia (No Intervention): Patients receiving "no intervention" will receive no intranasal ketamine while awaiting intravenous line placement for parenteral pain control.
- Intranasal Ketamine + Standard Analgesia (Active Comparator): Enrolled patients will receive one dose of Intranasal Ketamine dosed at 1mg/kg (Ketamine 500mg/10 mL solution) after triage while waiting for IV placement (max 50mg).
  Interventions: Drug: Intranasal ketamine

INTERVENTIONS:
Drug: Intranasal ketamine — Patients with vaso-occlusive episode and sickle cell disease in moderate to severe pain determined at triage will receive intranasal ketamine while awaiting IV placement.
  Arms: Intranasal Ketamine + Standard Analgesia

SUMMARY:
This will be a descriptive cohort study of intranasal ketamine as the initial analgesic for children with sickle cell disease who present to the pediatric emergency department with vaso-occlusive crisis and are awaiting intravenous line placement.

DETAILED DESCRIPTION:
This will be a prospective observational cohort involving patients 3 to 25 years of age who present to the Pediatric Emergency Department (PED) at Jacobi Medical Center with vaso-occlusive episode (VOE) in moderate-severe pain (FACES or numeric rating scale ≥5) as determined at triage. Currently, the standard of treatment for VOE at our institution is intravenous (IV) line placement and IV opioid analgesia. The patient will receive intranasal (IN) Ketamine as the first parental analgesic, so as to provide more immediate pain relief while they wait for IV placement and IV analgesia, for opioid pain control, which is currently the standard of care at our institution. The primary objective of this study is to describe the analgesic effect of IN ketamine in treating moderate-to-severe pain due to VOE in the pediatric ED as measured by a pain scale rating at various time intervals following administration. Secondary objectives are to describe the effect of IN ketamine on the need for additional doses of opioid medications, patient satisfaction and disposition.

ELIGIBILITY:
Inclusion Criteria:

* History of Hemoglobin SS or SC disease
* Age 3 years old to 25 years old presenting to the PED with vaso-occlusive with moderate-severe pain determined at triage as pain score (FACES or numeric rating scale) ≥ 5
* Parent or patient willing to provide consent/assent
* English speaking

Exclusion Criteria:

* Patient with concern for more severe complications including acute chest, splenic sequestration, sepsis, stroke, non-VOC pain, asthma exacerbation
* Allergy to ketamine
* GCS<15
* Obstructive nasal anatomy as per parent history
* History of a psychiatric disorder
* Pregnant patients will be excluded. Female patients > 12 years old are routinely tested for pregnancy in our PED. Patients found to be pregnant will not be enrolled in study.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score Using Wong Baker/FACES (age<11yr) | 30 minutes
  Change in pain rating from baseline to 30 minutes after initial administration of Ketamine. Pain assessments will be made using the Wong Baker FACES scale for children aged 10 years and younger. The Wong Baker/FACES scale is scored in multiples of 2 (each associated with a facial reaction), starting from a minimum of 0 to a maximum of 10.
Change in Pain Score Using Numeric Rating Scale (age>11yr) | 30 minutes
  Change in pain rating from baseline to 30 minutes after initial administration of Ketamine. For patients 11 yrs and older, pain will be assessed using the Numeric Rating Scale, which is a scale from a minimum of 0 to a maximum of 10.
Change in Pain Score Using Wong Baker/FACES (age<11yr) | 15 minutes
  Change in pain rating from baseline to 15 minutes after initial administration of Ketamine. Pain assessments will be made using the Wong Baker FACES scale for children aged 10 years and younger. The Wong Baker/FACES scale is scored in multiples of 2 (each associated with a facial reaction), starting from a minimum of 0 to a maximum of 10.
Change in Pain Score Using a Numeric Rating Scale (age>11yr) | 15 minutes
  Change in pain rating from baseline to 15 minutes after initial administration of Ketamine. For patients older than 11 years and older, pain will be assessed using the Numeric Rating Scale, which is a scale from a minimum of 0 to a maximum of 10.
Change in Pain Score Using Wong Baker/FACES (age<11yr) | 15 minutes
  Change in pain rating from baseline to 60 minutes after initial administration of Ketamine. Pain assessments will be made using the Wong Baker FACES scale for children aged 10 years and younger. The Wong Baker/FACES scale is scored in multiples of 2 (each associated with a facial reaction), starting from a minimum of 0 to a maximum of 10.
Change in Pain Score Using a Numeric Rating Scale (age>11yr) | 15 minutes
  Change in pain rating from baseline to 60 minutes after initial administration of Ketamine. For patients 11 years and older, pain will be assessed using the Numeric Rating Scale, which is a scale from a minimum of 0 to a maximum of 10.

SECONDARY OUTCOMES:
Additional Opiate Medication | Duration of ED visit, an average of 5 hrs
  Number of opiate analgesic doses and a comparison of opiate equivalents/kilogram versus mean dose for prior visits (if the patient has been seen for VOE prior)
Patient Satisfaction | At patient disposition, an average of 5 hrs
  Patient/Parent satisfaction based on questionnaire. Patients will answer based on a 4 point scale (not happy at all/a little happy/happy&satisfied/very happy)
Rate of Admission | Duration of ED visit, an average of 5 hrs
  Percentage of patients within each group who are admitted (vs discharged)
Rate of Return Visit | 1 week
  Percentage of patients within each group who have a return visit documented in the electronic medical record within 1 week of the ER visit.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jacobi Medical Center, The Bronx, New York
  - JACOBI, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No